CLINICAL TRIAL: NCT04530006
Title: Acetyl-Amantadine as a Biomarker in Patients With Glioblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CancerCare Manitoba (Other)
Collaborators: University of Manitoba (Other); The Metabolomics Innovation Centre (Unknown); BioMark Diagnostics Inc. (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 50604
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma Multiforme
Keywords: Acetyl-amantadine; GBM; Glioblastoma; Brain; diagnostic biomarker; MRI; tumor volume; amantadine; brain tumor; cancer patients
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients eligible for the study who have provided consent will be asked to ingest a regular 200mg dose of FDA approved drug Amantadine, according to timelines proposed in the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GBM Patients (Experimental): This cohort of patients will be asked to orally ingest 200mg dose of FDA approved drug amantadine hydrochloride. This will be done at the following timepoints:
  1. Within 4 weeks of the start of treatment; but as close to commencement of treatment (Day 1 of radiotherapy) as possible for newly diagnosed patients.
  2. Cycle 1, Day 1 of chemotherapy (temozolomide or lomustine) +/- 7 days
  3. Day 1 +/- 7 days for each visit where MRI is obtained (typically every 8-12 weeks - pre-cycles 4, 7, 10, for temozolomide or pre-cycles 3, 5, and 7 for lomustine)
  Interventions: Diagnostic Test: Amantadine Hydrochloride

INTERVENTIONS:
Diagnostic Test: Amantadine Hydrochloride — Patients who are eligible for the study will be administered a regular 200 mg dose of FDA approved drug amantadine. This will be done at the following timepoints:
  1. Within 4 weeks of the start of treatment; but as close to commencement of treatment (Day 1 of radiotherapy) as possible for newly diagnosed patients.
  2. Cycle 1, Day 1 of chemotherapy (temozolomide or lomustine) +/- 7 days
  3. Day 1 +/- 7 days for each visit where MRI is obtained (typically every 8-12 weeks - pre-cycles 4, 7, 10, for temozolomide or pre-cycles 3, 5, and 7 for lomustine)

SUMMARY:
Glioblastoma multiforme (GBM) is the most common brain tumor in adults. The strikingly poor survival for patients with GBM (average survival 14-16 months following diagnosis) is due in part to limited early detection methods and an absence of effective therapeutic options. The study proposed would establish important evidence for the use of Health Canada approved drugs such as amantadine as a safe, effective and affordable way to monitor GBM. The method is based on the overproduction of a key enzyme in GBM cells called spermine/ spermidine n-acetyl transferase (SSAT1). The increased SSAT1 expression in GBM results in increased metabolism of the drug which is detected in the blood or urine of patients with GBM. The levels of acetyl-amantadine captured will be correlated with the tumor burden as seen on the MRIs of these patients. Thus, the study aims to determine the usefulness of amantadine as a diagnostic biomarker for GBM.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common malignant primary brain tumor in adults, with a median age of onset of 55 to 60 years. Most patients are treated with postoperative radiation and chemotherapy following their initial surgery. For newly diagnosed, high grade gliomas, the first post-radiation cycle of temozolomide (an oral chemotherapy drug) typically begins four weeks after completion of radiation therapy1. During radiation, temozolomide or lomustine is given daily (seven days per week). Assessment of response and progression is made through brain magnetic resonance imaging (MRI) with contrast, which is typically obtained within one month after completion of radiation therapy and then every two months during adjuvant temozolomide to assess disease status1. With the available standard of care, the median overall survival of patients with glioblastoma remains very low - approximately 10 to 12 months2.

The poor prognosis with GBM is a result of an absence of early detection and ineffective treatment options. The proposed exploratory pilot project attempts to addresses the problem of accurate tumor progression monitoring in GBM through the development of a drug biomarker that monitors spermidine/spermine N1-acetyltransferase (SSAT1) activity. SSAT1 is an important enzyme involved in polyamine regulation in the cell. As polyamines are essential for tumor proliferation, SSAT1 is over-expressed in many different cancers, as shown in a number of non-clinical trials3,4,5. These trials provide a rationale for our project: if SSAT1 is overexpressed in cancers including glioblastoma, then a substrate of SSAT1 could serve as a biomarker for determining the cellular activity of SSAT1. An effective substrate is amantadine, and following its acetylation by SSAT1, N-acetyl-amantadine levels excreted in the blood and urine samples of patients with glioblastoma could be used to indicate the presence of upregulation of SSAT1, and therefore, indicative of cancer. Recently published clinical trials involving investigators here at University of Manitoba and CancerCare Manitoba have reported a method for assessing tumor progression in lung and breast cancer patients based on acetyl- amantadine levels in blood and urine6,7,8. The assay is predicated on the selective acetylation of the drug amantadine by SSAT1. Published studies indicate increases in acetyl-amantadine in blood and urine from patients receiving a single oral dose of amantadine was predictive of tumor burden. Tappia et.al.7 reported that human cancer is associated with high urinary concentration of acetyl-amantadine with receiver-operating characteristic (ROC) for acetyl-amantadine demonstrated to be 0.689 (CI: 0.591-0.786, 95%) in lung cancer and 0.717 (CI: 0.577-0.858, 95%) for breast cancer.

Given the use of acetyl-amantadine as an early biomarker for lung and breast cancer, the present study protocol examines the extent to which acetyl-amantadine levels in blood and urine can be used to detect glioblastoma progression, particularly tumor recurrence which happens in the majority of patients and is considered inevitable after a median survival time of 32 - 36 weeks1. There are currently no studies that have attempted to determine the diagnostic value of acetyl-amantadine in glioblastoma patients, and therefore, this would be a pilot project. Under this protocol, patients diagnosed with glioblastoma (newly or recurrent) who are following the standard of care (surgical resection and radiation/chemotherapy) will be enrolled in the study. An initial assessment of the participant's baseline acetyl-amantadine levels in blood will be determined at the first visit. Thereafter, participants will be administered a standard 200 mg dose of the Health Canada approved drug amantadine at every visit in which MRI based imaging assessments are being performed (typically, every 8 - 12 weeks). Blood and urine samples will be taken at each visit to assay for acetyl-amantadine levels. These resulting acetyl-amantadine levels will be correlated with MRI based image findings to determine the extent to which this biomarker can be used for treatment monitoring in glioblastoma patients.

While the hypothesis is that acetyl-amantadine levels in blood or urine can be used to track tumor progression, an increase in acetyl-amantadine level would not indicate per se what type of tumor was present. For this reason, a metabolic profile on blood and urine samples collected from glioblastoma patients will be performed, to determine if there is a metabolic signature that can be established for glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years+)
* Pathologically confirmed Glioblastoma
* ECOG performance status 0-2
* Planned treatment with radiation and/or chemotherapy with temozolomide or lomustine
* Able to return to the study centre for study visits
* Able to swallow oral pills
* Serum creatinine and creatinine clearance (>60mL/min)
* Liver enzymes for liver function (Liver function tests <2.5 times the upper limit of normal)
* Participants of childbearing potential must agree to use an effective contraceptive method.

Exclusion Criteria:

* Known hypersensitivity or allergy to amantadine
* Concurrent infection requiring antiviral medication
* Concurrent medication with known interaction with amantadine (see below)
* Previous diagnosis of Parkinson's disease or parkinsonism
* Previous diagnosis of schizophrenia
* Current use of methamphetamine or cocaine
* Inability to swallow oral pills
* Significant impairment in renal function (Creatinine clearance < 60 mL/min)
* Women who are pregnant or are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Blood and Urine Acetyl-Amantadine levels in patients with GBM | This outcome will be assessed every 8 to 12 weeks. This will continue through study completion, an average of two years.
  Samples of plasma and urine will be analyzed by established analytical methods (as developed by Biopharmaceutical Research Inc., Vancouver, B.C.; Health Canada and FDA approved). Quantitative analysis of amantadine and acetyl-amantadine in plasma and urine samples will be performed using liquid chromatography triple quadrupole tandem mass spectroscopy (LC-MS/MS). Samples (50 µl) will be spiked with 50 µl of internal standard, deuterated acetyl-amantadine (d3-Ac-amantidine), and proteins precipitated with 0.5 ml of ice-cold methanol. The lyophilized deproteinated samples are reconstituted in 0.1 ml of 0.1% formic acid. Samples are injected onto a C-18 stationary column and eluted using a gradient mobile phase consisting of 0.1% aqueous formic acid (A) and 0.1% formic acid in methanol (B). The run time for each sample is 9 minutes with the mobile phase starting at 5% B and increasing to 95% B during sample elution.

SECONDARY OUTCOMES:
GBM tumor volume in correlation with serum and urine acetyl-amantadine levels in patients with GBM | This outcome will be assessed every 8 to 12 weeks. This will continue through study completion, an average of two years.
  Standard of care MRI will be used. Definitions of response to standard therapy (progression, stable disease, response) will follow the established Response Assessment in Neuro-Oncology (RANO) guidelines9.
  Post-hoc volumetric analysis will be done using quantitative semi-automated Olea Sphere software (Olea Medical, France).
  The study does not require additional MRI scans to be performed; Routine MRI images, as per glioblastoma standard of treatment, are posted to Radiology Information System/Picture Archiving and Communication System (RISPACS) and will be accessed for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrom QT, Gittleman H, Xu J, Kromer C, Wolinsky Y, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2009-2013. Neuro Oncol. 2016 Oct 1;18(suppl_5):v1-v75. doi: 10.1093/neuonc/now207. No abstract available. PMID 28475809
- [Background] Babbar N, Hacker A, Huang Y, Casero RA Jr. Tumor necrosis factor alpha induces spermidine/spermine N1-acetyltransferase through nuclear factor kappaB in non-small cell lung cancer cells. J Biol Chem. 2006 Aug 25;281(34):24182-92. doi: 10.1074/jbc.M601871200. Epub 2006 Jun 6. PMID 16757480
- [Background] Gabrielson E, Tully E, Hacker A, Pegg AE, Davidson NE, Casero RA Jr. Induction of spermidine/spermine N1-acetyltransferase in breast cancer tissues treated with the polyamine analogue N1, N11-diethylnorspermine. Cancer Chemother Pharmacol. 2004 Aug;54(2):122-6. doi: 10.1007/s00280-004-0786-1. Epub 2004 May 8. PMID 15138709
- [Background] Huang W, Eickhoff JC, Mehraein-Ghomi F, Church DR, Wilding G, Basu HS. Expression of spermidine/spermine N(1) -acetyl transferase (SSAT) in human prostate tissues is related to prostate cancer progression and metastasis. Prostate. 2015 Aug 1;75(11):1150-9. doi: 10.1002/pros.22996. Epub 2015 Apr 20. PMID 25893668
- [Background] Tappia PS, Maksymiuk AW, Sitar DS, Akhtar PS, Khatun N, Parveen R, Ahmed R, Ahmed RB, Cheng B, Huang G, Bach H, Hiebert B, Ramjiawan B. Predictive value and clinical significance of increased SSAT-1 activity in healthy adults. Future Sci OA. 2019 Jul 1;5(7):FSO400. doi: 10.2144/fsoa-2019-0023. PMID 31428447
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676